CLINICAL TRIAL: NCT07300670
Title: The Effect of Losartan on Cephalexin
Acronym: KEFALOS
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aleksi Tornio (Other Government)
Collaborators: Turku University Hospital (Other Government); University of Turku (Other); University of Helsinki (Other); Helsinki University Central Hospital (Other)
Responsible Party: Sponsor-Investigator, Aleksi Tornio, Chief Physician, Turku University Hospital
Organization: Turku University Hospital (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KEFALOS
Record Dates: First submitted 2025-11-27; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Possible Interaction Between Losartan and Cephalexin; Healthy
Keywords: losartan; cephalexin; pharmacokinetic interaction; absorption
MeSH Terms: interventions — Losartan; Cephalexin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Sequence A (Other): water at 7.30, cephalexin 500 mg at 10.30; then water at 7.30, losartan 100 mg and cephalexin 500 mg at 10.30; then losartan 100 mg at 7.30, cephalexin 500 mg at 10.30
  Interventions: Drug: losartan; Drug: cephalexin
- Sequence B (Other): water at 7.30, losartan 100 mg and cephalexin 500 mg at 10.30; then water at 7.30, cephalexin 500 mg at 10.30; then losartan 100 mg at 7.30, cephalexin 500 mg at 10.30
  Interventions: Drug: losartan; Drug: cephalexin
- Sequence C (Other): losartan 100 mg at 7.30, cephalexin 500 mg at 10.30; then water at 7.30, losartan 100 mg and cephalexin 500 mg at 10.30; then water at 7.30, cephalexin 500 mg at 10.30
  Interventions: Drug: losartan; Drug: cephalexin
- Sequence D (Other): water at 7.30, cephalexin 500 mg at 10.30; then losartan 100 mg at 7.30, cephalexin 500 mg at 10.30; then water at 7.30, losartan 100 mg and cephalexin 500 mg at 10.30
  Interventions: Drug: losartan; Drug: cephalexin
- Sequence E (Other): water at 7.30, losartan 100 mg and cephalexin 500 mg at 10.30; then losartan 100 mg at 7.30, cephalexin 500 mg at 10.30; then water at 7.30, cephalexin 500 mg at 10.30
  Interventions: Drug: losartan; Drug: cephalexin
- Sequence F (Other): losartan 100 mg at 7.30, cephalexin 500 mg at 10.30; then water at 7.30, cephalexin 500 mg at 10.30; then water at 7.30, losartan 100 mg and cephalexin 500 mg at 10.30
  Interventions: Drug: losartan; Drug: cephalexin

INTERVENTIONS:
Drug: losartan — 100 mg tablet orally, single dose
  Other Names: Cozaar
Drug: cephalexin — 500 mg tablet orally, single dose
  Other Names: Kefalex; Kefexin

SUMMARY:
The goal of this clinical trial is to investigate the effects of the blood pressure-lowering drug losartan on the blood levels and urinary excretion of the antibiotic cephalexin during simultaneous and staggered ingestion in healthy volunteers. The main questions it aims to answer are:

1. Does losartan affect cephalexin levels and excretion when ingested at the same time?
2. Does a three-hour interval between ingestion of losartan and cephalexin eliminate a possible effect?

Researchers will compare the effects of losartan ingested at the same time, losartan ingested three hours prior, and no losartan ingested on oral cephalexin in each participant to see whether an interaction exists and could be avoided.

Participants will visit the research laboratory on three days during which they will ingest single doses of losartan at the same time with, three hours prior to, and not at all prior to ingesting single doses of cephalexin.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* 18-40 years of age
* good health
* systolic blood pressure of at least 115 mmHg
* all screening laboratory results (P-Krea, Pt-GFReEPI, P-Na, P-K, P-ALAT, P-AFOS, P-GT, B-PVK+T) acceptable; minor deviations from reference ranges are acceptable at the discretion of a physician-scientist with the exceptions of P-Krea and P-K which must be at or below the higher reference limit, and Pt-GFReEPI which must be at or above the reference limit (Reference limits: Tyks Laboratories, Turku University Hospital)
* regarding female subjects, a negative pregnancy test (S-HCG-O) before the study, and the use of an acceptable contraceptive method (e.g. condom, copper intrauterine device or abstinence from heterosexual intercourse), according to CTFG Recommendations related to contraception and pregnancy testing in clinical trials, are required

Exclusion Criteria:

* inability to provide written informed consent in Finnish
* remarkable illness
* confirmed or reasonably suspected allergy to cephalexin, amoxicillin, benzylpenicillin, phenoxymethylpenicillin, piperacillin, cefaclor, or cefamandole
* confirmed or reasonably suspected severe delayed allergic reaction to any beta-lactam antibiotic
* underweight (BMI less than 18.5 kg/m2)
* obesity (BMI greater than 30 kg/m2)
* smoking
* regular medication, including hormonal contraception in the form of pills, intrauterine device, subdermal implant etc.
* current or planned pregnancy, and breastfeeding
* less than three months elapsed since a prior clinical trial
* less than three months elapsed since donating blood

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Plasma concentrations of cephalexin over time, the cumulative urinary excretion of cephalexin, and the pharmacokinetic parameters derived from these measurements following simultaneous or staggered ingestion of losartan | up to 8 hours after ingestion of cephalexin on three consecutive days separated by at least one-week intervals

SECONDARY OUTCOMES:
Plasma concentrations of losartan and losartan carboxylic acid over time, the cumulative urinary excretion of losartan and losartan carboxylic acid, and the pharmacokinetic parameters derived from these measurements | up to 11 hours after ingestion of losartan or water on three consecutive days separated by at least one-week intervals
  following simultaneous and staggered ingestion of cephalexin

OTHER OUTCOMES:
Plasma and urinary concentrations of endogenous and diet-derived metabolites, and the effects of genetic variants and other individual factors on the pharmacokinetic parameters of cephalexin and losartan | up to 11½ hours on three consecutive days separated by at least one-week intervals

CONTACTS AND LOCATIONS:
Overall Officials: Aleksi Tornio, M.D., Ph.D., Principal Investigator — Unit of Clinical Pharmacology, Turku University Hospital
Locations (1):
- Unit of Clinical Pharmacology, Turku University Hospital, Turku, Southwest Finland, Finland

IPD SHARING:
Plan to Share IPD: No
The individual data supporting the findings of this study cannot be made available to other researchers to protect the privacy of the study subjects in accordance with European legislation and ethical requirements.